CLINICAL TRIAL: NCT03363945
Title: A Phase 3, Randomized, Multi-center, Open-label, Controlled Trial to Assess the Efficacy and Safety of Cellular Immunotherapy With MDR-101 for Induction of Immune Tolerance in Recipients of HLA-matched, Living Donor Kidney Transplants
Brief Title: Cellular Immunotherapy in Recipients of HLA-matched, Living Donor Kidney Transplants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medeor Therapeutics, Inc. (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MDR-101-MLK
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Kidney Transplant Rejection
Keywords: kidney transplant; cellular therapy; anti-rejection therapy; living donor; HLA-matched; hematopoietic stem cells (HSC); CD34+; CD3+; T cells

STUDY DESIGN:
Intervention Model Description: Total lymphoid irradiation and anti-thymocyte globulin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MDR-101 (Active Comparator): A single dose will be administered via IV infusion post-kidney transplant.
  Interventions: Biological: MDR-101
- Control Arm (No Intervention): Subjects randomized to this arm will receive the standard anti-rejection medications that would be given to kidney transplant recipients who are outside the study.

INTERVENTIONS:
Biological: MDR-101 — Enriched CD34+ hematopoietic stem cells and defined dose of CD3+ T-cells
  Arms: MDR-101

SUMMARY:
The primary objective of this study is to demonstrate the safety and efficacy of cellular immunotherapy with MDR-101 for induction of functional immune tolerance in recipients of human leukocyte antigen (HLA)-matched, living donor kidney transplants.

DETAILED DESCRIPTION:
Currently, patients receiving a transplanted kidney are required to take life-long immunosuppressive medications to prevent rejection of the transplanted kidney. These medications carry substantial side effects. In addition, these medicines often do not completely control damage to the kidney from the recipients' immune system, ultimately causing the kidney to fail.

Medeor Therapeutics is developing a novel cell-based therapy to reprogram the recipients' immune system to accept a transplanted kidney without the need for long term use of immunosuppression drugs.

The purpose of the current Phase 3 study is to demonstrate the efficacy and safety of MDR-101 for the induction of transplant immune tolerance in a prospective, randomized, multicenter clinical trial. MDR-101 is intended to induce mixed lymphohematopoietic chimerism and donor specific immune tolerance in order to preserve transplant kidney function, avert transplant kidney rejection, and eliminate the cumulative and serious side effects associated with immunosuppressive drugs.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Planned recipient of a first kidney allograft from an HLA-matched, living related donor
* Age ≥18 and ≤70 years
* Single solid organ recipient (kidney only)
* ABO matched with donor

Recipient Exclusion Criteria:

* Underlying kidney disease with a high risk of disease recurrence in the transplanted kidney
* Baseline positive donor-specific anti-HLA antibody testing
* Is taking immunosuppressive therapy
* Evidence of prior hepatitis B (HBV) or hepatitis C (HCV)

Donor Inclusion Criteria:

* HLA-matched first degree (parent, child or sibling) or second-degree (child of a sibling or half sibling) relative of the prospective recipient participant
* Age ≥18 and ≤70 years
* Prepared to be a living related kidney donor, and capable of undergoing G-CSF mobilization and apheresis of hematopoietic cells

Donor Exclusion Criteria:

* History of autoimmune disorders
* History of type 1 or type 2 diabetes mellitus
* Tests confirmed positive for human immunodeficiency virus (HIV), HBV, HCV, T. cruzi, or syphilis
* History of infection with Zika virus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Functional immune tolerance defined as | Up to 36 months post-kidney transplant
  * Achievement of the required duration of persistent donor mixed chimerism to permit calcineurin inhibitor immunosuppressive withdrawal beginning at 6-7 months post-kidney transplant surgery, and
  * Successful withdrawal from all immunosuppressives by at least 12 months post-kidney transplant surgery, and
  * Subsequent successful maintenance off all immunosuppressive drugs for at least 24 additional months (out to at least 36 months post-kidney transplant surgery) without biopsy-proven acute rejection, de novo Donor Specific Antibody, transplant kidney loss, or subject death. Loss to follow-up will be adjudicated as a failure in intent-to-treat analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Lenuta Micsa, MD, Study Director — Medeor Therapeutics
Locations (19):
- United States (18):
  - Loma Linda University Medical Center, Loma Linda, California
  - USC, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic Hospital, Jacksonville, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - RWJBarnabas Health, Orange, New Jersey
  - Upstate University Hospital, Syracuse, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - Intermountain Transplant Center, Murray, Utah
  - INOVA Fairfax Hospital, Fairfax, Virginia
  - University of Wisconsin School of Medicine, Madison, Wisconsin
- CIUSSS de l'Est- de-l'Île-de-Montréal Installation Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided